CLINICAL TRIAL: NCT04449016
Title: Effect of Ethnicity on Changes in VO2max and Cardiac Output in Response to Short-Term High Intensity Interval Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, San Marcos (Other)
Responsible Party: Principal Investigator, Todd A. Astorino Ph.D, PhD, FACSM, California State University, San Marcos
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 1200680-2
Record Dates: First submitted 2020-06-24; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Improved VO2max and Cardiac Output in Response to Training
Keywords: HIIT; Inactive; Women
MeSH Terms: conditions — Sedentary Behavior | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: This study was a longitudinal, repeated measures between subjects design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caucasian (Experimental): Participants performed 9 sessions of HIIT over 3 weeks, utilizing progressive overload by increasing the number of bouts by 1 each week. They started with 8 bouts on week 1, 9 bouts on week 2, and 10 bouts on week 3.
  Interventions: Other: High intensity interval training
- Hispanic (Experimental): Participants performed 9 sessions of HIIT over 3 weeks, utilizing progressive overload by increasing the number of bouts by 1 each week. They started with 8 bouts on week 1, 9 bouts on week 2, and 10 bouts on week 3.
  Interventions: Other: High intensity interval training

INTERVENTIONS:
Other: High intensity interval training — Repeated, brief, and intense exercise bouts separated by active recovery

SUMMARY:
The purpose of this study was to determine if ethnicity alters training responsiveness to a low dose of high intensity interval training in inactive women.

DETAILED DESCRIPTION:
Prior to the session, women completed a 4-minute warmup at 10 % PPO. Each subject completed 9 sessions of HIIT over a 3-week period which consisted of eight to ten 1-minute bouts of cycling at 85% PPO with 75-second recovery between bouts at 10 % PPO. This protocol is well-tolerated in inactive individuals. Continuously during each session, heart rate was monitored using telemetry. On days 1, 3, 6, and 9 of training, the physical activity enjoyment scale (PACES) was completed. VO2max and cardiac output max were assessed prior to training, as well as post.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Between the age of 18-45
* Healthy and non-obese (BMI < 30 kg/m2)
* Perform less than 150 minutes per week of exercise in the last 12 months
* 100% Caucasian or 100% Hispanic

Exclusion Criteria:

* Injured
* Obese
* Active
* Mixed ethnicity

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Change in baseline in VO2max at 3 weeks | 3 weeks
  Each participant performed VO2max testing on an electronically-braked cycle ergometer using a ramp protocol. During exercise, subjects expired through a plastic mouthpiece and low resistance valve into tubing connected to a mixing chamber. Measures of ventilation and expired fractions of oxygen and carbon dioxide were obtained throughout exercise by a metabolic cart. Gas exchange data including VO2, VCO2, and ventilation were time-averaged every 15 seconds. The test was terminated when the subject's pedal cadence was below 50 rev/min.
Change in baseline in cardiac output max at 3 weeks | 3 weeks
  During the VO2max assessment, participants wore a thoracic impedance device to measure heart rate and stroke volume, calculating their cardiac output.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Astorino, PhD, Principal Investigator — California State University, San Marcos
Locations (1):
- California State University San Marcos, San Marcos, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Raleigh JP, Giles MD, Scribbans TD, Edgett BA, Sawula LJ, Bonafiglia JT, Graham RB, Gurd BJ. The impact of work-matched interval training on V̇O2peak and V̇O2 kinetics: diminishing returns with increasing intensity. Appl Physiol Nutr Metab. 2016 Jul;41(7):706-13. doi: 10.1139/apnm-2015-0614. Epub 2016 Feb 29. PMID 27337599
- [Background] Astorino TA, White AC, Dalleck LC. Supramaximal testing to confirm attainment of VO2max in sedentary men and women. Int J Sports Med. 2009 Apr;30(4):279-84. doi: 10.1055/s-0028-1104588. Epub 2009 Feb 6. PMID 19199208
- [Background] Astorino TA, Schubert MM, Palumbo E, Stirling D, McMillan DW, Cooper C, Godinez J, Martinez D, Gallant R. Magnitude and time course of changes in maximal oxygen uptake in response to distinct regimens of chronic interval training in sedentary women. Eur J Appl Physiol. 2013 Sep;113(9):2361-9. doi: 10.1007/s00421-013-2672-1. Epub 2013 Jun 11. PMID 23754097
- [Background] Bowdon M, Marcovitz P, Jain SK, Boura J, Liroff KG, Franklin BA. Exercise Training in "At-Risk" Black and White Women: A Comparative Cohort Analyses. Med Sci Sports Exerc. 2018 Jul;50(7):1350-1356. doi: 10.1249/MSS.0000000000001580. PMID 29462100
- [Background] Gill JM, Celis-Morales CA, Ghouri N. Physical activity, ethnicity and cardio-metabolic health: does one size fit all? Atherosclerosis. 2014 Feb;232(2):319-33. doi: 10.1016/j.atherosclerosis.2013.11.039. Epub 2013 Nov 23. PMID 24468145
- [Background] Johnson JL, Slentz CA, Duscha BD, Samsa GP, McCartney JS, Houmard JA, Kraus WE. Gender and racial differences in lipoprotein subclass distributions: the STRRIDE study. Atherosclerosis. 2004 Oct;176(2):371-7. doi: 10.1016/j.atherosclerosis.2004.05.018. PMID 15380461
- [Background] Skinner JS, Jaskolski A, Jaskolska A, Krasnoff J, Gagnon J, Leon AS, Rao DC, Wilmore JH, Bouchard C; HERITAGE Family Study. Age, sex, race, initial fitness, and response to training: the HERITAGE Family Study. J Appl Physiol (1985). 2001 May;90(5):1770-6. doi: 10.1152/jappl.2001.90.5.1770. PMID 11299267